CLINICAL TRIAL: NCT05342727
Title: The Impact of Transcranial Direct and Alternating Stimulation of the Prefrontal Cortex at Different Intensities and Frequencies on Cognition of Schizophrenic Patients
Brief Title: Transcranial Direct and Alternating Stimulation of the Prefrontal Cortex for Cognitive Improvement in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Ardabil University of Medical Sciences (Other); Leibniz Research Centre for Working Environment and Human Factors (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, The National Brain Mapping Laboratory (NBML)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IR.ARUMS.REC.1400.043
Record Dates: First submitted 2022-03-26; First posted 2022-04-25 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia; Cognitive Dysfunction
Keywords: schizophrenia; tDCS; tACS; Cognition; dorsolateral prefrontal cortex
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel group and each group with crossover design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation Concealment is used to perform a random sequence on study participants. Also, non-transparent envelopes sealed with random sequences will be used, in a way that each random sequence is recorded on a card, and the cards are placed in the envelope in order. In order to maintain a random sequence, the envelopes are numbered in the same way on the outer surface. Finally, the lids of the envelopes are glued and placed inside a box. At the beginning of the registration, according to the order of entry of the eligible participants, one of the envelopes will be opened in order and the assigned group of the participant will be revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Active Comparator): The tDCS arm receives two real (or active) stimulation at 2 mA and 3 mA intensities and one placebo electrical stimulation for 20 minutes.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- tACS group (Active Comparator): The tACS arm receives two real (or active) stimulation at 8 Hz and 40 Hz frequencies and one placebo alternating electrical stimulation for 20 minutes.
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — In tDCS, direct electrical currents at the intensity of interest (2 mA for example) are generated by an electrical stimulator and are noninvasively delivered to the scalp through a pair of saline-soaked sponge electrodes (7×5 cm).
  Arms: tDCS group
Device: transcranial alternating current stimulation (tACS) — In tACS, alternating electrical currents at the frequency of interest (8 Hz for example) are generated by an electrical stimulator and are noninvasively delivered to the scalp through a pair of saline-soaked sponge electrodes (7×5 cm).
  Arms: tACS group

SUMMARY:
The purpose of this study is to investigate different stimulation intensities and frequencies of transcranial direct and alternating current stimulation over the dorsolateral prefrontal cortex for cognitive improvement in schizophrenia.

DETAILED DESCRIPTION:
In this randomized, double-blind study, 50 patients diagnosed with schizophrenia are randomly assigned into two arms. The first group receives transcranial direct current stimulation (tDCS) at three intensities (2 mA, 3 mA, and sham) and the second group receives transcranial alternating current stimulation (tACS) at three different frequencies (8 Hz, 40 Hz, and sham) over the left dorsolateral prefrontal cortex for 20 min. There are at least 72 hours between stimulation sessions. The patients conduct three cognitive tasks from the CANTAB neuropsychological battery for schizophrenia during stimulation including a working memory task, a cognitive flexibility task, and an emotion recognition task. Mood stability is also evaluated before and after each stimulation session with the Positive and Negative Affect Scale (PANAS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia based on DSM V,
* Being 18-50 years old (male and female)
* If female, negative urine pregnancy test
* feasibility for tDCS interventions according to safety guidelines
* stable medication regime especially the classical neuroleptics and all CNS-activating medications, if taken, 4-6 weeks before the experiment
* fluency in the native language
* right-handed
* Required written informed consent signed by patients' guardian

Exclusion Criteria:

* pregnancy
* alcohol or substance dependence
* history of seizure
* history of neurological disorder
* history of head injury
* Presence of ferromagnetic objects in the body that are contraindicated for brain stimulation of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Spatial Working Memory behavioral performance | During procedure (4 minutes)
  The test begins with a number of coloured squares (boxes) shown on the screen. The aim of this test is that by selecting the boxes and using a process of elimination, the participant should find one yellow 'token' in each of a number of boxes and use them to fill up an empty column on the right-hand side of the screen.
executive function behavioral performance | During procedure (8-10 minutes)
  The participant is shown two displays containing three coloured balls. The test administrator first demonstrates to the participant how to move the balls in the lower display to copy the pattern in the upper display and completes one demonstration problem, where the solution requires one move. The participant must then complete three further problems, one each requiring two moves, three moves and four moves. Next the participant is shown further problems and must work out in their head how many moves the solutions require and then select the appropriate box at the bottom of the screen to indicate their response
Emotional recognition behavioral performance | During procedure (60 minutes)
  Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200 milliseconds and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise)

SECONDARY OUTCOMES:
The Positive and Negative Affect Schedule (PANAS) | through study completion in each experimental session up to 1 hour
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Locations (1):
- Ardabil University of Medical Sciences, Ardabil, Iran

IPD SHARING:
Plan to Share IPD: No
Data will be available upon reasonable request from the PI after publication of results